CLINICAL TRIAL: NCT06216171
Title: Prospective Randomized Study on Adaptive Radiotherapy in Head and Neck Tumor Patients (Pro- Head and Neck -ART, ProHEART)
Brief Title: Adaptive Radiotherapy in Head and Neck Tumor Patients
Acronym: ProHEART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Maja Guberina, PD Dr. med. (MD) M. Guberina (senior consultant, specialist), University Hospital, Essen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 23-11674-BO
Record Dates: First submitted 2023-12-30; First posted 2024-01-22 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Head and Neck Neoplasms; Head and Neck Cancer; Adaptive Radiotherapy; Optimization
Keywords: Head and Neck Neoplasms; Head and Neck Cancer; Adaptive Radiotherapy; Optimization
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy, Image-Guided

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Adaptive Radiotherapy (Experimental): Adaptive Radiotherapy, online onboard adaptation of the dosis to actual anatomy of the day by a specialist of radiation oncology and a medical physicist
  Interventions: Radiation: Adaptive Radiotherapy
- Standard conventional Treatment Arm, IGRT (Active Comparator): Standard treatment option, image guided radiotherapy without online adaptation
  Interventions: Radiation: image guided radiotherapy without online adaptation

INTERVENTIONS:
Radiation: Adaptive Radiotherapy — Adaptive Radiotherapy
  Arms: Adaptive Radiotherapy
Radiation: image guided radiotherapy without online adaptation — image guided radiotherapy without online adaptation
  Arms: Standard conventional Treatment Arm, IGRT

SUMMARY:
Most newly diagnosed oropharyngeal and hypopharyngeal cancers are treated with radiochemotherapy with curative intent. If the field-set UP margins are broad, the consequence may be that quality of life is impaired. The study group of Nutting et al. (2023) investigated this year whether dysphagia-optimized intensity-modulated radiotherapy can reduce the radiation dose to structures associated with dysphagia and aspiration and improve swallowing function compared to standard IMRT (Nutting C, Finneran L, Roe J, Petkar I, Rooney K, Hall E; DARS Triallist Group. Dysphagia-optimized intensity-modulated radiotherapy versus standard radiotherapy in patients with pharyngeal cancer - Authors' reply. Lancet Oncol. 2023 Oct;24(10):e398. doi: 10.1016/S1470-2045(23)00457-6. PMID: 37797636.) The study group concluded that the results suggest that dysphagia-optimized IMRT improves patient-reported swallowing function compared to standard IMRT. DO-IMRT should be considered the new standard of care for patients receiving radiotherapy for pharyngeal cancer, and ART could further improve outcomes.

DETAILED DESCRIPTION:
Most newly diagnosed oropharyngeal and hypopharyngeal cancers are treated with radiochemotherapy with curative intent. If the field-set UP margins are broad, the consequence may be that quality of life is impaired. The study group of Nutting et al. (2023) investigated this year whether dysphagia-optimized intensity-modulated radiotherapy can reduce the radiation dose to structures associated with dysphagia and aspiration and improve swallowing function compared to standard IMRT (Nutting C, Finneran L, Roe J, Petkar I, Rooney K, Hall E; DARS Triallist Group. Dysphagia-optimized intensity-modulated radiotherapy versus standard radiotherapy in patients with pharyngeal cancer - Authors' reply. Lancet Oncol. 2023 Oct;24(10):e398. doi: 10.1016/S1470-2045(23)00457-6. PMID: 37797636.) The study group concluded that the results suggest that dysphagia-optimized IMRT improves patient-reported swallowing function compared to standard IMRT. DO-IMRT should be considered the new standard of care for patients receiving radiotherapy for pharyngeal cancer, and ART could further improve outcomes.

Thus, in this trial we analyze ART in head and neck cancer in a prospective randomized trial.

ELIGIBILITY:
Inclusion Criteria:

ECOG 0/1 No prior cancer treatment

Exclusion Criteria:

ECOG 2-4 Prior cancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
EORTC CTC AE Score | 2 months - 5 years
  quality of life, Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 Published: November 27, 2017
Dysphagia score | 2 months - 5 years
  Dysphagia score

SECONDARY OUTCOMES:
Overall Survival | 2-5 years
  Overall Survival
Progression Free Survival | 2-5 years
  Progression Free Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Maja Guberina, Essen, Germany

IPD SHARING:
Plan to Share IPD: No